CLINICAL TRIAL: NCT01336257
Title: Effectiveness of a Decision Support System in Improving the Diagnosis and Screening Rate of Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Italiano de Buenos Aires (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Damian Borbolla, MD, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HIBA00019
Record Dates: First submitted 2011-04-14; First posted 2011-04-15 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Breast Cancer
Keywords: Decision Support Techniques; Electronic Health Records; Reminder Systems; Early Detection of Cancer; Mammography; Women
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electronic Reminder (Experimental): alert from SEBASTIAN decision support system
  Interventions: Other: SEBASTIAN Clinical Decision Support System (CDSS)
- control (No Intervention)

INTERVENTIONS:
Other: SEBASTIAN Clinical Decision Support System (CDSS) — SEBASTIAN is an example of a clinical decision support technology that supports the latest, service-based architectural approach to CDSS implementation. Developed at Duke University, SEBASTIAN is a clinical decision support Web service whose interface is now the basis of the HL7 Decision Support Service draft standard SEBASTIAN places a standardized interface in front of clinical decision support knowledge modules and makes only limited demands on how relevant patient data are collected or on how decision support inferences are communicated to end-users
  Arms: Electronic Reminder

SUMMARY:
Clinical decision support has been shown to improve the performance of screening tests; however, few studies have documented direct clinical benefit resulting from the increased screening promoted by clinical decision support systems.

The purpose of this study was to determine if a standards-based, sophisticated decision support system could not only promote additional breast cancer screening, but also detect significantly more breast cancer

DETAILED DESCRIPTION:
Breast cancer is the most common female cancer. In the United States, the second most common cause of cancer death in women, and the main cause of death in women ages 45 to 55 years old. The U.S. Preventive Services Task Force recommends screening mammography, with or without clinical breast examination, every one to two years among women aged 50 to 69 years old.

Recent research has shown that health care delivered in industrialized nations often falls short of optimal, evidence based care. US adults receive only about half of recommended care. To address these deficiencies in care, health-care organizations are increasingly turning to clinical decision support systems. A clinical decision-support system is any computer program designed to help health-care professionals to make clinical decisions. In a sense, any computer system that deals with clinical data or knowledge is intended to provide decision support.

Examples include manual or computer based systems that attach care reminders to the charts of patients needing specific preventive care services and computerized physician order entry systems that provide patient-specific recommendations as part of the order entry process. Such systems have been shown to improve prescribing practices, reduce serious medication errors, enhance the delivery of preventive care services, and improve adherence to recommended care standards.

The aim of this study is to show the efficacy of a decision-support system as a strategy for improving the performance of the mammography care process and the detection of significantly more breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women between 50 and 69 years old

Exclusion Criteria:

* Breast Neoplasms
* Bilateral mastectomy
* Disabled Persons

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with new Breast Neoplasms Diagnosis (Incident cases) | 18 month
  New Breast Neoplasms Diagnosis (Incident cases from biopsy reports). Breast Neoplasms are stored in the institutional Clinical Data Repository. The diagnosis are automatically codified using a terminology server that use SNOMED-CT as reference terminology

SECONDARY OUTCOMES:
Number of patient with breast cancer screening due that received the order to perform the study (mammography) | 18 month
  Number of patient with breast cancer screening due that received the order to perform the study (mammography). This information will be record through the clinical data repository every time that a provider order a screening test to each of the patients involve in the study

CONTACTS AND LOCATIONS:
Overall Officials: Damian A Borbolla, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires, Argentina